CLINICAL TRIAL: NCT00003093
Title: Treatment for Infants and Children With Intermediate Risk Neuroblastoma: A Phase III Intergroup CCG/POG Study
Brief Title: Combination Chemotherapy in Treating Children With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3961; COG-A3961 (Other: Children's Oncology Group); CCG-A3961 (Other: Children's Cancer Group); POG-A3961 (Other: Pediatric Oncology Group); CDR0000065804 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Biological: sargramostim; Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen®; NSC #614629
Biological: sargramostim
  Other Names: Granulocyte Macrophage-Colony Stimulating Factor; rhu GM-CSF; GM-CSF; Prokine; Leukine; NSC #613795
Drug: carboplatin
  Other Names: Paraplatin; NSC-241240
Drug: cyclophosphamide
  Other Names: Cytoxan; NSC-26271
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC-123127
Drug: etoposide
  Other Names: VP-16; VePesid; NSC-141540
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Combination chemotherapy plus surgery may be an effective treatment for neuroblastoma.

PURPOSE: This phase III trial is studying how well combination chemotherapy followed by surgery works in treating young patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the use of selected prognostic variables to assign treatment increases the event-free survival and overall survival in children with intermediate-risk neuroblastoma.
* Determine the acute and long-term morbidity and toxicity of surgery and combination chemotherapy in this patient population.
* Assess the relationship between extent of tumor resection and event-free and overall survival in patients treated with this regimen.

OUTLINE: Patients receive carboplatin IV over 1 hour on days 0, 21, and 63; cyclophosphamide IV over 1 hour on days 21 and 42; doxorubicin IV over 15-60 minutes on days 21 and 63; and etoposide IV over 2 hours on days 0-2, 42-44, and 63-65. Patients under 60 days of age also receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning 24 hours after the last chemotherapy administration and continuing until blood counts recover. Patients with favorable biology who do not achieve complete remission then undergo surgery to remove or debulk residual disease on day 84 or when blood counts recover. Patients with favorable biology who achieve partial response and surgery to the primary site is not deemed in the best interest of the patient may receive additional chemotherapy (as below) and delay surgery to the primary site after completion of chemotherapy.

Patients with unfavorable biology receive additional chemotherapy comprising cyclophosphamide IV over 1 hour on days 84, 105, and 147; etoposide IV over 2 hours on days 84-86 and 126-128; carboplatin IV over 1 hour on days 105 and 126; and doxorubicin IV over 15-60 minutes on days 105 and 147. Patients then undergo debulking surgery on day 168 or when blood counts recover.

Some patients may then undergo radiotherapy after surgery.

Patients are followed monthly for 6 months, every 2 months for 6 months, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven neuroblastoma or maturing ganglioneuroma that is judged to be intermediate risk by one of the following criteria:

  * International Neuroblastoma Staging System (INSS) stage III

    * Under 1 year old, MYCN oncogene nonamplified, and any ploidy
    * 1 to 20 years old, MYCN nonamplified, favorable Shimada histology
  * INSS stage IV

    * Under 1 year old, MYCN nonamplified, any ploidy
  * INSS stage IVS

    * Under 1 year old, MYCN nonamplified, unfavorable Shimada histology and any ploidy OR favorable Shimada histology and diploidy
* All patients must be registered on the companion neuroblastoma biology study (COG-ANBL00B1)

PATIENT CHARACTERISTICS:

Age:

* Under 21

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No abnormal organ function that would prohibit chemotherapy unless due to neuroblastoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy for patients with intradural extension and emergent paresis allowed provided biopsy was performed within 96 hours after treatment

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other prior therapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 573 (Actual)
Dates: Start 1988-03; Primary Completion 2006-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: David L. Baker, MD, MBBS, FRACP, FRCPA, Study Chair — Princess Margaret Hospital for Children
Locations (235):
- United States (207):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Children's Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Pediatric Specialty Clinic at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis/St. Paul, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Children's Hospital at Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cancer Center at Baylor College of Medicine, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- University Medical Center Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Children's Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Dubois SG, Geier E, Batra V, Yee SW, Neuhaus J, Segal M, Martinez D, Pawel B, Yanik G, Naranjo A, London WB, Kreissman S, Baker D, Attiyeh E, Hogarty MD, Maris JM, Giacomini K, Matthay KK. Evaluation of Norepinephrine Transporter Expression and Metaiodobenzylguanidine Avidity in Neuroblastoma: A Report from the Children's Oncology Group. Int J Mol Imaging. 2012;2012:250834. doi: 10.1155/2012/250834. Epub 2012 Sep 25. PMID 23050139
- [Background] Marachelian A, Shimada H, Sano H, Jackson H, Stein J, Sposto R, Matthay KK, Baker D, Villablanca JG. The significance of serial histopathology in a residual mass for outcome of intermediate risk stage 3 neuroblastoma. Pediatr Blood Cancer. 2012 May;58(5):675-81. doi: 10.1002/pbc.23250. PMID 22493777
- [Background] Meany HJ, Attiyeh EF, Naranjo A, et al.: Outcome analysis of non-high-risk neuroblastoma patients enrolled on Children's Oncology Group trials P9641 and A3961. [Abstract] J Clin Oncol 30 (Suppl 15): A-9533, 2012.
- [Background] Attiyeh EF, Mosse YP, Diskin S, et al.: Identification of genomic DNA signatures predicting relapse in low- and intermediate- risk neuroblastoma using a case control design and high-density SNP genotyping: a Children's Oncology Group (COG) study. [Abstract] J Clin Oncol 25 (Suppl 18): A-9500, 526s, 2007.
- [Result] Baker DL, Schmidt ML, Cohn SL, Maris JM, London WB, Buxton A, Stram D, Castleberry RP, Shimada H, Sandler A, Shamberger RC, Look AT, Reynolds CP, Seeger RC, Matthay KK; Children's Oncology Group. Outcome after reduced chemotherapy for intermediate-risk neuroblastoma. N Engl J Med. 2010 Sep 30;363(14):1313-23. doi: 10.1056/NEJMoa1001527. PMID 20879880
- [Result] Baker DL, Schmidt M, Cohn S, et al.: A phase III trial of biologically-based therapy reduction for intermediate risk neuroblastoma. [Abstract] J Clin Oncol 25 (Suppl 18): A-9504, 2007.